CLINICAL TRIAL: NCT03060824
Title: Changes in Plasma Osmolality Related to the Use of Cardiopulmonary Bypass With Hyperosmolar Prime, an Observational Study.
Brief Title: Changes in Plasma Osmolality Related to the Use of Cardiopulmonary Bypass With Hyperosmolar Prime.
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/509-31
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-03

CONDITIONS: Cardiopulmonary Bypass
Keywords: Osmolality; Sodium; CABG; Cardiovascular Diseases; Cardiopulmonary bypass
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG with the aid of CPB.: Cardiac surgical patients subjected to coronary artery bypass grafting with the aid of Cardiopulmonary Bypass. Perioperative measurements of osmolality in plasma.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — To explore changes in osmolality during coronary artery bypass grafting surgery with the aid of Cardiopulmonary Bypass by repeated measurements of osmolality and concentration shifts of sodium, glucose and urea in plasma.

SUMMARY:
During the use of Cardiopulmonary Bypass (CPB) for cardiac surgery there is an instant mixture of the patient's blood and the fluid needed to fill the extracorporeal circuit before use. This will change the composition of the body fluids. This study aims to plot these changes in regard to particle concentration (osmolality).

DETAILED DESCRIPTION:
During the use of CPB for cardiac surgery there is an instant mixture of the patient's blood and the fluid needed to prime the extracorporeal circuit. Many studies have pointed to the benefits of using a hyperosmolar prime to counteract formation of tissue oedema. Rapid changes in osmolality may as a serious consequence lead to osmotic demyelination syndrome. At the Heart Centre of Umeå University Hospital, Sweden, there is a tradition of using a hyperosmolar prime. This study aims to explore changes in osmolality during coronary artery bypass grafting surgery by repeated measurements of osmolality and concentration shifts of sodium, glucose and urea in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 yr
* New York Heart Association Functional Classification(NYHA) I-III
* Body Surface Area(BSA) 1.8-2.5 m2

Exclusion Criteria:

* Diabetes
* Estimated Glomerular Filtration Rate(eGFR)<50ml/min/1,73 m2

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to coronary artery bypass grafting with the aid of Cardiopulmonary Bypass.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Changes in plasma osmolality | Before surgery; repeated during surgery and on postoperative day 1 and 2.
  Repeated measurements of plasma osmolality aim to outline changes in plasma osmolality related to the use of hyperosmolar prime.

SECONDARY OUTCOMES:
Change in osmolar gap | Before surgery; repeated during surgery and on postoperative day 1 and 2.
  Analysing urea, sodium and glucose in plasma using the same sampling intervals as for plasma osmolality enables calculation of the osmolar gap and to set its relation to the use of hyperosmolar prime

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Hedström, MD, Principal Investigator — Heart Centre, Umeå University Hospital, Sweden
Locations (1):
- Heart Centre, Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after reviewing final results after study completion at this site and through publication in a scientific journal.

REFERENCES:
- [Background] Gu YJ, Boonstra PW. Selection of priming solutions for cardiopulmonary bypass in adults. Multimed Man Cardiothorac Surg. 2006 Jan 1;2006(109):mmcts.2005.001198. doi: 10.1510/mmcts.2005.001198. PMID 24415398
- [Background] Giuliani C, Peri A. Effects of Hyponatremia on the Brain. J Clin Med. 2014 Oct 28;3(4):1163-77. doi: 10.3390/jcm3041163. PMID 26237597
- [Derived] Malmqvist G, Claesson Lingehall H, Appelblad M, Svenmarker S. Cardiopulmonary bypass prime composition: beyond crystalloids versus colloids. Perfusion. 2019 Mar;34(2):130-135. doi: 10.1177/0267659118793249. Epub 2018 Aug 16. PMID 30114960
- [Derived] Drury NE, Horsburgh A, Bi R, Willetts RG, Jones TJ. Cardioplegia practice in paediatric cardiac surgery: a UK & Ireland survey. Perfusion. 2019 Mar;34(2):125-129. doi: 10.1177/0267659118794343. Epub 2018 Aug 10. PMID 30095360